CLINICAL TRIAL: NCT02375074
Title: Supported Employment and Preventing Early Disability (SEED)
Brief Title: Supported Employment and Preventing Early Disability
Acronym: SEED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NORCE Norwegian Research Centre AS (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 227002/H20
Record Dates: First submitted 2014-12-03; First posted 2015-03-02 (Estimated); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Unemployment
Keywords: Supported Employment; Vocational Rehabilitation; Youth; Sick leave; Disability; Coping; Work; Occupational; Labor market participation; Randomized Controlled Trial
MeSH Terms: interventions — Employment, Supported

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supported Employment (Experimental): Supported Employment (SE), focusing on competitive employment in real-life settings without long-lasting preceding training.
  Interventions: Behavioral: Supported Employment
- Traditional Vocational Rehabilitation (Experimental): Traditional Vocational Rehabilitation (TVR), offering training and preparation for the labor market in a sheltered environment.
  Interventions: Behavioral: Traditional Vocational Rehabilitation

INTERVENTIONS:
Behavioral: Supported Employment — Supported Employment (SE), focusing on competitive employment in real-life settings without long-lasting preceding training.
  Arms: Supported Employment
Behavioral: Traditional Vocational Rehabilitation — Traditional Vocational Rehabilitation (TVR), offering training and preparation for the labor market in a sheltered environment
  Arms: Traditional Vocational Rehabilitation

SUMMARY:
The share of young workers falling into early work disability is an increasingly important problem in Norway. Early withdrawal or exclusion from the labor market leads to large individual and societal costs. The SEED-trial is a randomized controlled trial aiming to provide evidence-based knowledge about different approaches to prevent permanent disability and increase labor market participation in this important and vulnerable group. The trial includes young adults aged 18-30 years who are at risk of early work disability, and the participants will be randomly assigned to 1 of 2 interventions, both aimed at facilitating participation in working life:

1. Traditional Vocational Rehabilitation (TVR), offering training and preparation for the labor market in a sheltered environment
2. Supported Employment (SE), focusing on competitive employment in real-life settings without long-lasting preceding training

Both interventions are currently provided by The Norwegian Labor and Welfare Administration (NAV). Supported Employment was introduced recently and is currently being implemented, while traditional vocational rehabilitation with sheltered employment has been around for years. However, no Norwegian controlled studies have been conducted on these practices in this population. The current study will therefore provide new knowledge of the effect of traditional as well as new and promising interventions to increase labor market participation and prevent early disability.

DETAILED DESCRIPTION:
A detailed study protocol was published in BMC Public Health in 2016, and is openly available in fulltext at: https://bmcpublichealth.biomedcentral.com/articles/10.1186/s12889-016-3280-x

ELIGIBILITY:
Inclusion criteria:

* Not in employment or education
* Receiving temporary benefits
* Intended for the VR service "traineeships in sheltered businesses"

Exclusion criteria:

* Not expressing interest in getting help to obtain competitive work
* Insufficient language skills to answer questionnaires in Norwegian

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2014-05; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Any competitive employment (yes/no) | 12 months
  Several sources of information for competitive employment will be used: Survey data for hours worked and success in employment, and register data for receipt of social security benefits, income, financial assistance, and educational activity.

SECONDARY OUTCOMES:
Physical and mental health | 12 months
  Survey data (anxiety, depression, disability, fatigue, subjective health complaints, quality of life)
Coping | 12 months
  Survey data
Illness perceptions | 12 months
  Survey data
Alcohol and drug abuse | 12 months
  Survey data
Cost effectiveness | 12 months
  Cost/benefit analysis

CONTACTS AND LOCATIONS:
Overall Officials: Silje Endresen Reme, PhD, Principal Investigator — NORCE Norwegian Research Centre
Locations (1):
- NORCE Norwegian Research Centre, Bergen, Norway

REFERENCES:
- [Result] Sveinsdottir V, Lie SA, Bond GR, Eriksen HR, Tveito TH, Grasdal AL, Reme SE. Individual placement and support for young adults at risk of early work disability (the SEED trial). A randomized controlled trial. Scand J Work Environ Health. 2020 Jan 1;46(1):50-59. doi: 10.5271/sjweh.3837. Epub 2019 Jun 6. PMID 31170299
- [Derived] Sveinsdottir V, Eriksen HR, Baste V, Hetland J, Reme SE. Young adults at risk of early work disability: who are they? BMC Public Health. 2018 Oct 16;18(1):1176. doi: 10.1186/s12889-018-6095-0. PMID 30326872
- [Derived] Sveinsdottir V, Tveito TH, Bond GR, Grasdal AL, Lie SA, Reme SE. Protocol for the SEED-trial: Supported Employment and preventing Early Disability. BMC Public Health. 2016 Jul 15;16:579. doi: 10.1186/s12889-016-3280-x. PMID 27422271